CLINICAL TRIAL: NCT04536857
Title: Detection of A-synuclein Aggregate as Biomarker in Diagnosing Parkinson's Disease at Early Stage by Using Protein Misfolding Cyclic Amplification (PMCA)
Status: Withdrawn | Type: Observational
Why Stopped: Our applied project did not receive funding support, so it cannot proceed, leading to the withdrawal of the study.
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jian Wang, Professor & Deputy Director, Department of Neurology, Huashan Hospital
Other Study IDs: 2020 Provisional Audit No.1004
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease (PD); αSyn aggregates; Protein misfolding cyclic amplification (PMCA); Early diagnosis; CSF
MeSH Terms: conditions — Parkinson Disease; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Parkinson's Disease: Subjects who have a PD diagnosis
  Interventions: Other: Biomarker assay
- Multiple System Atrophy: Subjects who have an MSA diagnosis
  Interventions: Other: Biomarker assay
- Progressive Superanuclear Palsy: Subjects who have a PSP diagnosis
  Interventions: Other: Biomarker assay
- Age-matched controls: Subjects who do not have a diagnosed neurological disorder
  Interventions: Other: Biomarker assay

INTERVENTIONS:
Other: Biomarker assay — Biomarker assay will be used to quantify levels of misfolded alpha-synuclein aggregates in cerebrospinal fluid from patients with Parkinson's disease, multiple system atrophy, progressive superanuclear palsy and controls.

SUMMARY:
The study will investigate the biomarker of a-synuclein aggregate in CSF detected by protein misfolding cyclic amplification (PMCA) and its sensitivity and specificity in diagnosing Parkinson's disease at H-Y stage I and disease duration less than 1 year, compared with that from age-matched controls without neurodegeneration, those with Multiple System Atrophy (MSA) as a disease control with a-synucleinopathy, and those with Progressive Supranuclear Palsy (PSP) as a control with non-a-synucleinopathy neurodegeneration.

DETAILED DESCRIPTION:
This will be an observational study aiming to develop the protein misfolding cyclic amplification (PMCA) technology that detects minute amounts of αSyn aggregates circulating in cerebrospinal fluid (CSF) as a novel assay with high sensitivity and specificity for the early diagnosis of PD. To achieve this goal, we will apply the PMCA to detect the αSyn aggregates in the CSF samples acquired from a discovery cohort that consist of well-characterized early PD patients (disease duration ≤1 year and Hoehn and Yahr Stage I, and DAT-PET and FDG-PET meet the imaging features of PD, n=75) and gender, age-matched healthy controls (n=38). Furthermore, we will confirm the findings in a separate confirmatory cohort with well-characterized early PD patients (disease duration ≤1 year and Hoehn and Yahr Stage I, and DAT-PET and FDG-PET meet the imaging features of PD, n=75), early multiple system atrophy (MSA) patients (disease duration ≤1 year, n=38), early progressive supranuclear palsy (PSP) patients (disease duration ≤1 year, n=38) and age-matched healthy controls (n=38). The sensitivity, specificity, positive predictive value, negative predictive value, and area under curve of the PMCA for the early diagnosis of PD will be calculated in the discovery cohort and be confirmed in the confirmatory cohort, respectively. In addition, the clinical characteristics, including motor and nonmotor symptoms of early PD, MSA and PSP patients in the two cohort will be comprehensively assessed at baseline and during followed-up. To assess the value of the PMCA technology in the evaluation of the disease severity and progress, we will perform the partial correlation analysis between clinical features of early PD patients and the PMCA T50 defined as the time needed to reach 50% of the maximum aggregation.

Misfolded αSyn aggregates have the potential to serve as a biomarker for early PD. The PMCA technology could detect small quantities of misfolded αSyn aggregates by taking advantage of their ability to nucleate further aggregation, enabling a very high amplification of the signal. This study examines the effectiveness of using the PMCA as a novel technique for discriminating early PD from gender, age-matched healthy controls and other early parkinsonian disorders (MSA, PSP) by detecting small misfolded αSyn aggregates in CSF.

ELIGIBILITY:
For early PD patients

Inclusion criteria:

* Clinical diagnosis of "probable PD" by two neurologists specializing in movement disorders according to the International Parkinson and Movement Disorder Society (MDS) Clinical Diagnostic Criteria for PD (2015);
* Age 50-75, disease duration is less than 1 year, and Hoehn & Yahr Stage I;
* the dopamine reuptake transporter (DAT) is significantly reduced in striatum on PET imaging;
* Metabolic brain network detected by fluorine-18-labelled-fluorodeoxyglucose-PET(18F-FDG PET) is consistent with Parkinson's disease-related pattern (PDRP), with FDG hypermetabolism being in basal ganglia and cerebellum;
* Good response to anti-PD medications;
* Ability of completing questionnaires;
* Ability of providing informed consent;
* Willingness of being assessed by neurologists during off-medication state defined as discontinuing anti-PD medications for at least 12 hours before assessment.

Exclusion criteria:

* Secondary parkinsonism (ie. drug induced);
* Atypical parkinsonisms like MSA or PSP etc;
* Presence of any item in 10 red flags of the MDS Clinical Diagnostic Criteria for PD (2015) in the comprehensive assessments during follow-up;
* History of being diagnosed as any cancer within 5 years;
* Presence of any condition risking the procedure of performing lumbar puncture (LP);
* Pregnancy;
* Inability to comply with study procedures.

For early MSA patients

Inclusion criteria:

* Clinical diagnosis of "probable MSA" by two neurologists specializing in movement disorders according to the International Parkinson and Movement Disorder Society (MDS) second consensus criteria for MSA (2019);
* Age 50-75, and disease duration is less than 1 year;
* Metabolic brain network detected by fluorine-18-labelled-fluorodeoxyglucose-PET(18F-FDG PET) is consistent with MSA related pattern;
* Ability of completing questionnaires;
* Ability of providing informed consent;
* Willingness of being assessed by neurologists during off-medication state defined as discontinuing anti-PD medications for at least 12 hours before assessment.

Exclusion criteria:

* Secondary parkinsonism (ie. drug induced);
* History of being diagnosed as any cancer within 5 years;
* Presence of any condition risking the procedure of performing lumbar puncture (LP);
* Pregnancy;
* Inability to comply with study procedures.

For PSP patients

Inclusion criteria:

* Clinical diagnosis of "probable PSP" by two neurologists specializing in movement disorders according to MDS Clinical Diagnostic Criteria for PSP (2017);
* Age 50-75, disease duration is less than 1 year;
* Metabolic brain network detected by fluorine-18-labelled-fluorodeoxyglucose-PET(18F-FDG PET) is consistent with PSP related pattern;
* Ability of completing questionnaires;
* Ability of providing informed consent;
* Willingness of being assessed by neurologists during off-medication state defined as discontinuing anti-PD medications for at least 12 hours before assessment.

Exclusion criteria:

* Secondary parkinsonism (ie. drug induced);
* History of being diagnosed as any cancer within 5 years;
* Presence of any condition risking the procedure of performing lumbar puncture (LP);
* Pregnancy;
* Inability to comply with study procedures.

For controls without diagnosis of neurodegenerative disorders

Inclusion criteria:

* Age 50-75;
* No history of neurodegenerative disease of the central nervous system;
* No history of infective disease of the central system;
* Ability of completing questionnaires;
* Ability of providing informed consent.

Exclusion criteria:

* With prodromal symptoms of PD, such as rapid eye movement sleep behavior disorder (RBD);
* History of being diagnosed as any cancer within 5 years;
* Presence of any condition increasing the risk of the procedure of performing lumbar puncture (LP);
* Pregnancy;
* Inability to comply with study procedures.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Discovery cohort: (1) Early PD patients (disease duration ≤1 year and Hoehn and Yahr Stage I, n=75); (2) Gender, age-matched healthy controls (n=38); (3) The dopamine reuptake transporter (DAT) is significantly reduced in striatum on PET imaging; (4) Metabolic brain network detected by fluorine-18-labelled-fluorodeoxyglucose-PET(18F-FDG PET) is consistent with Parkinson's disease-related pattern (PDRP).
  Confirmatory cohort: (1) Early PD patients (disease duration ≤1 year and Hoehn and Yahr Stage I, n=75); (2) Early Multiple System Atrophy (MSA) patients (disease duration ≤1 year, n=38); (3) Early progressive supranuclear palsy (PSP) patients (disease duration ≤1 year, n=38); (4) Gender, age-matched healthy controls (n=38); (5) The dopamine reuptake transporter (DAT) is significantly reduced in striatum on PET imaging; (6) Metabolic brain network detected by fluorine-18-labelled-fluorodeoxyglucose-PET(18F-FDG PET) is consistent with Parkinson's disease-related pattern (PDRP).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The area under curve of the PMCA for the early diagnosis of PD | two years
  The area under curve is used to show the ability of the a-syn-PMCA to diagnose early PD. The value of area under curve is higher, then the ability of the a-syn-PMCA to diagnose early PD is stronger.

SECONDARY OUTCOMES:
The correlation between the PMCA T50 and MDS-UPDRS III score at baseline in PD patients | two years
  PMCA T50 is the time needed to reach 50% of the maximum aggregation. The motor symptoms of PD patients will be assessed using the Movement Disorder Society-Unified Parkinson's Disease Rating Scale Part 3 (MDS-UPDRS- III).
The correlation between PMCA T50 and subregional DAT in striatum in PD patients | two years
  PMCA T50 is the time needed to reach 50% of the maximum aggregation. The DAT uptake value (caudate, anterior putamen and/or posterior putamen) will be quantified using DAT-PET.
The correlation between PMCA T50 and PDRP expression value in PD patients | two years
  PMCA T50 is the time needed to reach 50% of the maximum aggregation. The Parkinson's disease-related pattern (PDRP) expression value will be quantified by using FDG-PET.
The correlation between PMCA T50 and the change of MDS-UPDRS III score between the baseline and the follow-up | two years
  PMCA T50 is the time needed to reach 50% of the maximum aggregation. The change of MDS-UPDRS III score is the difference of that between the baseline and the follow-up.
The sensitivity | two years
  The sensitivity is used to show the ability of the a-syn-PMCA to diagnose early PD patients, and is represented by true positive/ (true positive +false negative).
The specificity | two years
  The specificity is used to show the ability of the a-syn-PMCA to avoid false early PD patients and rule out early PD patients, and is represented by true negative/ (false positive + true negative).
The positive predictive value | two years
  The positive predictive value is used to show the ability of the a-syn-PMCA to correctly label early PD patients who test positive, and is represented by true positive / (true positive + false positive).
The negative predictive value | two years
  The negative predictive value is used to show the ability of the a-syn-PMCA to correctly label people who test negative, and is represented by true negative / (false negative + true negative).

CONTACTS AND LOCATIONS:
Overall Officials: Jian Wang, MD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided